CLINICAL TRIAL: NCT02142582
Title: Comparison of Different Oral Rehydration Solutions (ORS) in Short Bowel Syndrome (SBS) Patients on Home Parenteral Nutrition (HPN): A Prospective Double-blinded Randomized Controlled Trial.
Brief Title: Comparison of Different Oral Rehydration Solutions
Acronym: ORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13-008346
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Short Bowel Syndrome
Keywords: Home Parenteral Nutrition; Compliance; Short Bowel Syndrome; Oral Rehydration Solution
MeSH Terms: conditions — Short Bowel Syndrome; Patient Compliance; Osteoarthritis | interventions — World Health Organization oral rehydration solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- WHO ORS (Active Comparator): Participants will be instructed to dilute contents of the provided ORS to a 1 liter bottle and sip all day.
  Interventions: Dietary Supplement: WHO ORS
- Commercial ORS (Active Comparator): Participants will be instructed to dilute contents of the provided ORS to a 1 liter bottle and sip all day.
  Interventions: Dietary Supplement: Commercial ORS

INTERVENTIONS:
Dietary Supplement: WHO ORS — Participants will be randomized into one of the two groups. They will be provided with one of the two ORS solutions. Then, they will be followed for 6 months.
  Other Names: World Health Organization ORS
  Arms: WHO ORS
Dietary Supplement: Commercial ORS — Participants will be instructed to dilute contents of the provided ORS to a 1 liter bottle and sip all day.
  Other Names: Dripdrop
  Arms: Commercial ORS

SUMMARY:
Compliance is the biggest challenge in patients with Short Bowel Syndrome (SBS) on Home Parenteral Nutrition. These patients need to hydrate themselves to meet the excess fluid loss due to their anatomy. Oral Rehydration Solution (ORS) is prescribed to all these patients. The investigators believe that taste of the standard ORS is the biggest reason why these patients are not complaint. The new ORS in the market has been prepared with this in mind. The investigators want to study if this new ORS will improve the compliance in this patient cohort.

ELIGIBILITY:
Inclusion Criteria

* All patients with short bowel syndrome treated by the HPN program.

Exclusion Criteria

* Participants who have do not provide written consent.
* Participants who lack the ability to provide informed consent
* Participants who are not anticipated to be on HPN for at least 6 months (determined by PrincipaI Investigator).
* Pregnant women
* Participants with pre-existing congestive heart failure, acute/ chronic kidney failure. (determined by the PrincipaI Investigator)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients who will regularly take Oral Rehydration Solution (ORS) when the newly available ORS is compared to the World Health Organisation ORS. | 6 months

SECONDARY OUTCOMES:
Changes in the electrolytes in subjects using the commercial ORS versus the WHO ORS | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hurt, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States